CLINICAL TRIAL: NCT07031895
Title: Evaluation of the Efficacy of Xenograft Containing Hyaluronic Acid in Socket Preservation Procedure Radiologically and Histologically: A Prospective Randomized Controlled Clinical Study
Brief Title: The Effectiveness of Hyaluronic Acid in Bone Regeneration
Acronym: socket healing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Duygu Kilic, PhD, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/184-F
Record Dates: First submitted 2025-06-02; First posted 2025-06-22 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Socket Preservation
Keywords: Socket Preservation; hyaluronic acid; bone formation
MeSH Terms: interventions — Hyaluronic Acid; Transplantation, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bovine-derived graft/xenograft enriched with hyaluronic acid study group (Experimental): Study group - Patients whose alveolar bone is pre-evaluated using cone-beam computed tomography (CBCT) will receive a bovine-derived graft/xenograft enriched with hyaluronic acid in the extraction socket after tooth removal. Patients will be evaluated clinically, radiologically, and histologically at 4 months. Dental implants will be placed in the edentulous areas where the graft was applied. Bone samples will be collected during the preparation of the implant sockets and analyzed histologically. A third CBCT scan will be performed 6 months after implant placement to radiographically assess new bone formation and implant success.
  Interventions: Combination Product: a bovine-derived graft/xenograft enriched with hyaluronic acid
- Standard bovine-derived graft/xenograft comparison group (Active Comparator): Comparison group - Patients whose alveolar bone is pre-evaluated using CBCT will receive a standard bovine-derived graft/xenograft in the extraction socket after tooth removal. Patients will be evaluated clinically, radiologically, and histologically at 4 months. Dental implants will be placed in the grafted areas. Bone samples will be collected during implant socket preparation and analyzed histologically. A third CBCT scan will be performed 6 months after implant placement to assess new bone formation and implant success.
  Interventions: Combination Product: a standart bovine-derived graft/xenograft
- Control group without graft material (No Intervention): Control group - Patients whose alveolar bone is pre-evaluated using CBCT will undergo tooth extraction without graft material application, allowing for natural healing of the socket. Patients will be evaluated clinically, radiologically, and histologically at 4 months. Dental implants will be placed in the edentulous areas. Bone samples will be collected during the preparation of the implant sockets and analyzed histologically. A third CBCT scan will be performed 6 months after implant placement to assess new bone formation and implant success.

INTERVENTIONS:
Combination Product: a bovine-derived graft/xenograft enriched with hyaluronic acid — In study group a bovine-derived graft/xenograft enriched with hyaluronic acid will be placed in the extraction socket after tooth removal.
  Arms: Bovine-derived graft/xenograft enriched with hyaluronic acid study group
Combination Product: a standart bovine-derived graft/xenograft — In comparison group a standard bovine-derived graft/xenograft will be placed in the extraction socket after tooth removal.
  Arms: Standard bovine-derived graft/xenograft comparison group

SUMMARY:
Bone loss due to resorption is commonly observed in the alveolar socket following tooth extraction. This situation makes it difficult to preserve sufficient bone volume that would allow for ideal implant placement in cases requiring dental implants. Alveolar ridge preservation is a procedure aimed at minimizing bone resorption and preserving the volume and morphology of the alveolar ridge after tooth extraction.

The aim of this study is to evaluate the clinical effectiveness of socket preservation using a xenograft enriched with hyaluronic acid in patients with defective extraction sockets.

This study is designed as a randomized, controlled clinical trial including three parallel groups:

Study group - Patients whose alveolar bone was evaluated using cone-beam computed tomography (CBCT) will undergo tooth extraction, followed by the application of a bovine-derived graft/xenograft enriched with hyaluronic acid into the socket. Patients will be evaluated clinically, radiologically, and histologically at the 4th month. Dental implants will be placed in the edentulous areas where the graft was applied. Bone samples will be taken during the preparation of the implant sockets, and the bone tissue will be examined histologically. A third CBCT scan will be taken 6 months after implant placement to assess new bone formation and implant success radiographically.

Comparison group - Patients whose alveolar bone was evaluated using CBCT will undergo tooth extraction, followed by the application of a standard bovine-derived graft/xenograft into the socket. Patients will be evaluated clinically, radiologically, and histologically at the 4th month. Dental implants will be placed in the edentulous areas where the graft was applied. Bone samples will be taken during the preparation of the implant sockets, and the bone tissue will be examined histologically. A third CBCT scan will be taken 6 months after implant placement to assess new bone formation and implant success radiographically.

Control group - Patients whose alveolar bone was evaluated using CBCT will undergo tooth extraction, and the socket will be left to heal naturally without the application of any graft material. Patients will be evaluated clinically, radiologically, and histologically at the 4th month. Dental implants will be placed in the edentulous areas. Bone samples will be taken during the preparation of the implant sockets, and the bone tissue will be examined histologically. A third CBCT scan will be taken 6 months after implant placement to assess new bone formation and implant success radiographically.

DETAILED DESCRIPTION:
Following tooth extraction, volume loss due to bone resorption is observed in the alveolar socket. This condition complicates the preservation of sufficient bone volume that would allow for ideal implant placement in cases requiring dental implants. Alveolar ridge preservation is a procedure aimed at minimizing bone resorption and maintaining the volume and morphology of the alveolar ridge after tooth extraction. In this procedure, the goal is to provide structural support and a scaffold for new bone formation by using materials such as autogenous grafts, allografts, xenografts, barrier membranes, platelet-rich fibrin, bone morphogenetic proteins, and other growth factors. This approach supports bone regeneration by promoting osteogenesis and osteoconduction. Although current methods maintain their effectiveness, variability in outcomes is still observed. This highlights the need for more extensive research into different graft materials and innovative approaches.

Hyaluronic acid has emerged as a promising biomaterial for alveolar ridge preservation due to its multifaceted biological effects on tissue regeneration and wound healing. Its viscoelastic properties help maintain hydration and structural integrity at the graft site, reducing graft shrinkage and supporting vertical stability. Additionally, by interacting with cell surface receptors, it stimulates osteoblast activity and inhibits osteoclastogenesis, thereby contributing to increased bone density and improved biointegration of the graft material. Clinical studies have also demonstrated that hyaluronic acid enhances angiogenesis, strengthening the osteoconductive properties of graft materials and optimizing clinical outcomes in alveolar ridge preservation.

The aim of this study is to evaluate the clinical efficacy of socket preservation using a xenograft enriched with hyaluronic acid in patients with defective extraction sockets. Over a 10-month period, the study group receiving a hyaluronic acid-enriched xenograft will be compared with a control group receiving a standard xenograft and another control group left to natural healing after tooth extraction. Evaluated outcomes include horizontal and vertical bone gain, graft stability, residual graft, bone marrow presence, and bone mineral density.

This study is designed as a randomized, controlled clinical trial including three parallel groups:

Study group - Patients whose alveolar bone is pre-evaluated using cone-beam computed tomography (CBCT) will receive a bovine-derived graft/xenograft enriched with hyaluronic acid in the extraction socket after tooth removal. Patients will be evaluated clinically, radiologically, and histologically at 4 months. Dental implants will be placed in the edentulous areas where the graft was applied. Bone samples will be collected during the preparation of the implant sockets and analyzed histologically. A third CBCT scan will be performed 6 months after implant placement to radiographically assess new bone formation and implant success.

Comparison group - Patients whose alveolar bone is pre-evaluated using CBCT will receive a standard bovine-derived graft/xenograft in the extraction socket after tooth removal. Patients will be evaluated clinically, radiologically, and histologically at 4 months. Dental implants will be placed in the grafted areas. Bone samples will be collected during implant socket preparation and analyzed histologically. A third CBCT scan will be performed 6 months after implant placement to assess new bone formation and implant success.

Control group - Patients whose alveolar bone is pre-evaluated using CBCT will undergo tooth extraction without graft material application, allowing for natural healing of the socket. Patients will be evaluated clinically, radiologically, and histologically at 4 months. Dental implants will be placed in the edentulous areas. Bone samples will be collected during the preparation of the implant sockets and analyzed histologically. A third CBCT scan will be performed 6 months after implant placement to assess new bone formation and implant success.

Histopathological Studies Tissue samples collected for histological analysis will be fixed in 10% formaldehyde solution for 72 hours. After fixation, samples will undergo decalcification using a solution composed of 10% formaldehyde, 80% distilled water, and 10% nitric acid. Following decalcification, standard histological tissue processing will be performed. Prepared sections will be stained with Hematoxylin and Eosin (H&E) for general histological structure and Masson's Trichrome (MT) specifically for connective tissue evaluation. Microscopic evaluation will be performed using an Olympus BX51 light microscope (Olympus Corp., Tokyo, Japan) according to defined criteria, and measurements will be analyzed statistically using the ImageJ software program.

The obtained histological images will be evaluated according to Jerry Bouquot's classification (UTHSC School of Dentistry, Houston):

Grade 0 - No bone formation observed

Grade 1 - Minimal bone formation observed

Grade 2 - Moderate bone formation observed

Grade 3 - Considerable bone formation observed

Grade 4 - Extensive bone formation observed

Tissues collected from the study will also be analyzed using immunohistochemical staining to show the expression of Tartrate Resistant Acid Phosphatase (TRAP) and Alkaline Phosphatase (AP). For the different experimental groups, AP (Anti-Alkaline Phosphatase Antibody 100 μl, Abcam cat no: ab95462) will be used to demonstrate osteoblast activity, and TRAP (Rabbit Anti TRAP/Tartrate Resistant Acid Phosphatase Polyclonal Antibody, Bioss cat no: bs-6434R) will be used to determine osteoclast activity.

ImageJ software will be used at X40 magnification to calculate the intensity of AP and TRAP immunoreactivity in all femoral sections collected from the subjects in all experimental groups, and the results will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Socket type: Sockets with less than 50% bone resorption in the buccal and palatal/lingual walls according to the Kim JJ classification (Type I-IVa)

Age range: 18-65 years

Absence of active periodontal disease

No systemic diseases

Patients who will attend regular follow-up visits

Exclusion Criteria:

* Smoking

Uncontrolled systemic disease

Presence of infection in the area

Use of medications affecting bone metabolism

Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-02 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
bone formation | until the end of the histological examination 4 months after the socket preservation procedure
  At the 4-month follow-up, dental implants will be placed in the edentulous areas where grafts were applied. During the preparation of the implant sockets, bone samples will be collected and examined histologically.
  Tissue samples obtained for histological examination will be fixed in a 10% formaldehyde solution for 72 hours. Following fixation, the tissues will undergo a decalcification process. After decalcification, a routine histological tissue processing protocol will be applied.
  The obtained histological images will be evaluated according to the classification by Jerry Bouquot.
  Tissues obtained from the study will also be analyzed using immunohistochemical staining under a light microscope (Olympus BX51, Tokyo, Japan). The sections will be examined under a light microscope (Olympus BX51, Tokyo, Japan). For all femoral sections obtained from subjects in the experimental groups, the intensity of AP and TRAP immunoreactivity will be calculated at 40× magnification using the ImageJ.

SECONDARY OUTCOMES:
Radiographic bone evaluation | up to the radiographic evaluations at 4 and 10 months after the socket preservation procedure
  Cone-beam computed tomography (CBCT) scans will be obtained from each patient at three different time points throughout the study:
  Before socket preservation
  At 4 months after socket preservation (prior to implantation)
  At 6 months after implantation
  Using these scans, bone density, vertical and horizontal gain parameters will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Kılıç, PhD, Study Director — Erciyes University Faculty of Dentistry Department of Periodontology; Fidan Gulıyeva, Research Assistant, Principal Investigator — Erciyes University Faculty of Dentistry Department of Periodontology

IPD SHARING:
Plan to Share IPD: No
We do not wish to share data due to the possibility that patients may not consent to the sharing of personal information.

REFERENCES:
- [Background] Kloss FR, Kau T, Heimes D, Kammerer PW, Kloss-Brandstatter A. Enhanced alveolar ridge preservation with hyaluronic acid-enriched allografts: a comparative study of granular allografts with and without hyaluronic acid addition. Int J Implant Dent. 2024 Oct 9;10(1):42. doi: 10.1186/s40729-024-00559-6. PMID 39382763
- See also: Enhanced alveolar ridge preservation with hyaluronic acid-enriched allografts: a comparative study of granular allografts with and without hyaluronic acid addition — https://pubmed.ncbi.nlm.nih.gov/39382763/
- See also: Clinical and histologic outcomes of socket grafting after flapless tooth extraction: a systematic review of randomized controlled clinical trials — https://pubmed.ncbi.nlm.nih.gov/25749077/
- See also: Tissue changes of extraction sockets in humans: a comparison of spontaneous healing vs. ridge preservation with secondary soft tissue healing — https://pubmed.ncbi.nlm.nih.gov/22784417/